CLINICAL TRIAL: NCT04099901
Title: Anakinra: Efficacy of Anakinra for the Management of Fever During Neutropenia and Mucositis in Patients With Multiple Myeloma Receiving an Autologous Hematopoietic Stem Cell Transplantation After High-dose Melphalan - An RCT
Brief Title: Anakinra: Efficacy in the Management of Fever During Neutropenia and Mucositis in ASCT - A Randomized Controlled Trial
Acronym: AFFECT-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: University Medical Center Groningen (Other); Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HEMSC42
Record Dates: First submitted 2019-09-18; First posted 2019-09-23 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2023-11

CONDITIONS: Multiple Myeloma
Keywords: Anakinra; Mucositis; Hematopoietic stem cell transplantation; Febrile neutropenia
MeSH Terms: conditions — Multiple Myeloma; Mucositis; Febrile Neutropenia | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Intervention Model Description: Double-blind placebo-controlled randomized trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anakinra (Experimental): Dosage form: intravenous. Dosage: 300 mg. Frequency: once daily. Duration: 15 days (day -2 until day +12).
  Interventions: Drug: Anakinra
- Placebo (Placebo Comparator): Dosage form: intravenous. Dosage: not applicable. Frequency: once daily. Duration: 15 days (day -2 until day +12).
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Anakinra — Subjects will be treated with a daily dose of 300 mg anakinra, intravenously, starting on day -2, until day +12 (day 0 is day of SCT).
  Other Names: Kineret
  Arms: Anakinra
Drug: Placebos — Subjects will be treated with a daily dose of placebo, intravenously, starting on day -2, until day +12 (day 0 is day of SCT).
  Arms: Placebo

SUMMARY:
Oral and intestinal mucositis are major risk factors for the occurrence of fever during neutropenia and bloodstream infections after intensive chemo- and radiotherapy. These complications often require dose reductions or cause delay of treatment, and thereby interfere with optimal anticancer treatment. Currently, there are no effective strategies to prevent or treat mucositis and the related complications.

The pro-inflammatory cytokine interleukin-1β (IL-1β) has shown to be pivotal in the pathogenesis of mucositis and recently, it has been established in murine models that IL-1 inhibition significantly ameliorates chemotherapy-induced intestinal mucositis.

The investigators recently conducted a phase IIa study (AFFECT-1, NCT03233776) studying the safety and maximum tolerated dose of anakinra, a recombinant human IL-1 receptor antagonist in adult patients with multiple myeloma receiving high-dose melphalan (HDM) in the preparation for an autologous hematopoietic stem cell transplantation (ASCT) who are at high risk for experiencing mucositis and fever during neutropenia (FN).

Since treatment with anakinra has shown to be safe in this study population, the investigators will continue with a double-blind randomized placebo-controlled multicenter phase IIb trial to establish efficacy in the management of fever during neutropenia and mucositis.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Diagnosed with multiple myeloma
* Scheduled to receive an autologous SCT after myeloablative therapy with high-dose melphalan
* Managed with a central venous catheter (triple- or quadruple lumen)
* Is able and willing to participate
* Has provided written informed consent
* Has negative serology for active hepatitis B and C
* Has negative serology for HIV
* Has no known hypersensitivity to Escherichia coli derived products or any components of anakinra
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation (during treatment with study medication), and for 30 days after the last dose.

Exclusion Criteria:

* Inability to understand the nature and extent of the trial and the procedures required
* Enrollment in any other investigational treatment study or use of an investigational agent during the stem cell transplantation (this means studies in multiple myeloma regarding induction or maintenance treatment are permitted).
* Women who are pregnant or nursing
* Diagnosed with amyloidosis or light-chain deposition disease
* ALT or AST greater than 2.0 x upper limit of normal (ULN) of the local laboratories values.
* Bilirubin levels greater than 2.0 x upper limit of normal (ULN) of the local laboratories values, except for benign non-malignant indirect hyperbilirubinemia such as Gilbert syndrome
* Impaired renal function with eGFR <40 ml/min
* Received a live vaccine during the 3 months prior to baseline visit
* Recent use of IL-1 antagonist, such as anakinra, rilonacept or canakinumab, within three months prior to baseline visit
* Treatment with TNFα inhibiting agents (such as etanercept, adalimumab, infliximab, certolizumab and golimumab).
* Uncontrolled bacterial or viral infections, or fungal infections, at the start of therapy
* Colonization with methicillin-resistant Staphylococcus aureus (MRSA), carbapenemase-producing Enterobacteriaceae (CPE) or vancomycin-resistant enterococci (VRE) prior to registration
* Gram-negative colonization resistant to prophylaxis with ciprofloxacin or colistin/cotrimoxazole
* Subjects who are not able to receive antibacterial prophylaxis with ciprofloxacin or colistin/cotrimoxazole (because of hypersensitivity or drug interactions)
* Subjects with an active solid malignancy prior to registration, with the exception of cutaneous basal or squamous cell carcinomas
* History of mycobacterial infection.
* Subjects with intrinsic disorders of the gastro-intestinal (GI) tract, including, but not limited to: Crohn's disease, ulcerative colitis, celiac disease, short bowel syndrome.
* Subject has any concurrent medical or psychiatric condition or disease that is likely to interfere with the study procedures or results, or that in the opinion of the investigator, would constitute a hazard for participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
Reduction of the incidence of fever during neutropenia | Primary outcome will be determined during the period of hospitalization (day of admission [day -3] until discharge, maximum period +30 days).

SECONDARY OUTCOMES:
Reduction in incidence of mucositis-related fever | Outcome will be determined during the period of hospitalization (day of admission [day -3] until discharge, maximum period +30 days).
Daily mean CRP level | Outcome will be determined during the period of hospitalization (day of admission [day -3] until discharge, maximum period +30 days).
Intestinal mucositis as measured by the area-under-the-curve of reciprocal citrulline levels | Outcome will be determined during the period of hospitalization (day of admission [day -3] until discharge, maximum period +30 days).
Clinical mucositis as determined by the daily mouth and gut scores | Outcome will be determined during the period of hospitalization (day of admission [day -3] until discharge, maximum period +30 days).
Days with fever (≥ 38.5° C) | Outcome will be determined during the period of hospitalization (day of admission [day -3] until discharge, maximum period +30 days).
Incidence of bloodstream infections i.e. bacteremia | Outcome will be determined during the period of hospitalization (day of admission [day -3] until discharge, maximum period +30 days).
Length of hospital stay in days | Outcome will be determined during the period of hospitalization (day of admission [day -3] until discharge, maximum period +30 days).
Use of systemic antimicrobial agents (incidence and duration) | Outcome will be determined during the period of hospitalization (day of admission [day -3] until discharge, maximum period +30 days).
Use of analgesic drugs (incidence and duration) | Outcome will be determined during the period of hospitalization (day of admission [day -3] until discharge, maximum period +30 days).
Use of total parenteral nutrition (TPN) (incidence and duration) | Outcome will be determined during the period of hospitalization (day of admission [day -3] until discharge, maximum period +30 days).
Quality of life according to the EORTC QLQ-C30 | Baseline, +30 days/discharge (whichever comes first), +100 days, +1 year
  Quality of life according to the EORTC QLQ-C30
Fatigue severity according to the FACIT-Fatigue scale | Baseline, +30 days/discharge (whichever comes first), +100 days, +1 year
  Severity of fatigue as the score measured by the validated FACIT-Fatigue scale
Short term overall survival | +100 days and +1 year
Tumor response evaluation | +100 days and +1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Blijlevens, MD PhD, Principal Investigator — Radboud University Medical Center; Gerwin Huls, MD PhD, Principal Investigator — University Medical Center Groningen; Bart Biemond, MD PhD, Principal Investigator — Amsterdam UMC; Martijn Bakker, MD, Principal Investigator — University Medical Center Groningen
Locations (3):
- Netherlands (3):
  - Amsterdam UMC, location AMC, Amsterdam
  - University Medical Center Groningen (UMCG), Groningen
  - Radboudumc, Nijmegen

REFERENCES:
- [Derived] de Mooij CEM, van Groningen LFJ, de Haan AFJ, Biemond BJ, Bakker M, van der Velden WJFM, Blijlevens NMA. Anakinra: efficacy in the management of fever during neutropenia and mucositis in autologous stem cell transplantation (AFFECT-2)-study protocol for a multicenter randomized double-blind placebo-controlled trial. Trials. 2020 Nov 23;21(1):948. doi: 10.1186/s13063-020-04847-5. PMID 33225965